CLINICAL TRIAL: NCT05739916
Title: An Open Label, Randomized, Single Dose, Cross-over ,Two-group Study to Evaluate the Pharmacokinetics and Safety of DA-1229_01 5/1000mg in Healthy Subjects at Fed State
Brief Title: Phamacokinetics and Safety Profiles of DA-1229_01 5/1000mg in Healthy Subjects at Fed State
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 22-4250-BE025
Record Dates: First submitted 2023-02-13; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Healthy
MeSH Terms: interventions — Lead

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A(Before→ After) (Experimental)
  Interventions: Drug: DA-1229_01 5/1000mg (Before); Drug: DA-1229_01 5/1000mg (After)
- Sequence B(After→ Before) (Experimental)
  Interventions: Drug: DA-1229_01 5/1000mg (Before); Drug: DA-1229_01 5/1000mg (After)

INTERVENTIONS:
Drug: DA-1229_01 5/1000mg (Before) — single dose administration (one tablet once a day)
Drug: DA-1229_01 5/1000mg (After) — single dose administration (one tablet once a day)

SUMMARY:
This Phase I clinical study is to evaluate the safety/tolerability and pharmacokinetics of DA-1229_01(5/1000 mg x1 tablets) at fed state.

ELIGIBILITY:
Inclusive Criteria:

* Healthy Volunteers
* BMI between 18 and 30 kg/m2
* Body weight : Male≥50kg, Female≥45kg

Exclusion Criteria:

* Allergy or Drug hypersensitivity
* Clinically significant Medical History

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-03-30 (Estimated); Primary Completion 2023-04-28 (Estimated); Study Completion 2023-04-28 (Estimated)

PRIMARY OUTCOMES:
AUCt | pre-dose~48 hours post-dose
  area under the curve
Cmax | pre-dose~48 hours post-dose
  maximum plasma concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Metro Hospital, Anyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided